CLINICAL TRIAL: NCT06530927
Title: Micro-clots and Neutrophil Activation as Potential Indicators for Stroke Risk and Reperfusion Failure The CLOTSAFE - Study (Micro-CLOTs, Stroke Risk, Activated Neutrophils, Reperfusion FailurE)
Brief Title: Microclots and Neutrophil Activation as Potential Indicators for Stroke Risk and Reperfusion Failure
Acronym: CLOTSAFE
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Empa, Swiss Federal Laboratories for Materials Science and Technology (Other)
Responsible Party: Principal Investigator, Susanne Wegener, Prof. Dr. med., University of Zurich
Other Study IDs: 2024-01353
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke
Keywords: microclots; activated neutrophils; reperfusion failure; 3D rotational digital tomography
MeSH Terms: conditions — Ischemic Stroke | interventions — Microscopy, Atomic Force

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Control Group: Patients without previous documented stroke
  Interventions: Diagnostic Test: 3D rotational digital tomography; Diagnostic Test: Atomic Force Microscopy
- Chronic Stroke Group: Patients with previous stroke ≥1year ago
  Interventions: Diagnostic Test: 3D rotational digital tomography; Diagnostic Test: Atomic Force Microscopy
- Acute Stroke No Therapy Group: Patients with acute stroke, but without intravenous thrombolysis or mechanical thrombectomy
  Interventions: Diagnostic Test: 3D rotational digital tomography; Diagnostic Test: Atomic Force Microscopy
- Acute Stroke IVT only Group: Patients with acute stroke and intravenous thrombolysis
  Interventions: Diagnostic Test: 3D rotational digital tomography; Diagnostic Test: Atomic Force Microscopy
- Acute Stroke MT-Group: Patients with acute stroke and mechanical thrombectomy
  Interventions: Diagnostic Test: 3D rotational digital tomography; Diagnostic Test: Atomic Force Microscopy; Diagnostic Test: Micro-Computertomography

INTERVENTIONS:
Diagnostic Test: 3D rotational digital tomography — DHTM is label-free and records the phase shift of low-energy light passing through the specimen on a transparent surface with minimal perturbation. DHTM measures the refractive index (RI) and computes the refractive index gradient (RIG), unveiling optical heterogeneity in cells. We will analyze blood samples for the detection of altered neutrophil phenotypes and microclots.
Diagnostic Test: Atomic Force Microscopy — The atomic force microscope (AFM) is widely used in materials science and has found many applications in biological sciences but has been limited in use in vision science. The AFM can be used to image the topography of soft biological materials in their native environments. We will analyze blood samples for the detection of altered neutrophil phenotypes and microclots
Diagnostic Test: Micro-Computertomography — Micro-CT is a 3D imaging technique utilizing X-rays to see inside an object, slice by slice. Micro-CT, also called microtomography or micro computed tomography, is similar to hospital CT or "CAT" scan imaging but on a small scale with greatly increased resolution. Samples can be imaged with pixel sizes as small as 100 nanometers and objects can be scanned as large as 200 millimeters in diameter. We will use micro-CT to analyze blood clots from patients with large vessel occlusion.
  Groups: Acute Stroke MT-Group

SUMMARY:
Stroke remains a major health burden worldwide. Many patients are severely disabled and stay in need of care. Mechanical thrombectomy has dramatically improved outcomes for stroke patients with large vessel occlusions, yet 40-50% of patients with successful recanalization remain severely disabled despite successful recanalization, a scenario called "futile recanalization". One of the causes for this lack of treatment effect is capillary obstruction, or "no reflow", potentially resulting from activated neutrophils and micrometer-sized blood clots. To address this issue, we employ digital holotomographic and atomic force microscopy to investigate the structural and chemical characteristics of blood and clot material in stroke patients and individuals at high risk of developing a stroke. Our study elucidates the association of activated neutrophils and microclots with stroke risk, and may be associated with clinical outcome, stroke ethology and reperfusion failure in patients with stroke. Leveraging label-free microscopy tools, could potentially lead to the discovery of new biomarkers for individualized stroke treatment and prevention, ultimately offering rapid identification of at risk patients and improving clinical outcomes

DETAILED DESCRIPTION:
Background:

Stroke remains a major health burden worldwide. Many patients are severely disabled and stay in need of care. Since introducing mechanical thrombectomy as a therapeutic option, clinical outcome has drastically improved over the last few years. However, despite successful macrovascular reperfusion (recanalization), patients with stroke still have a significant risk (about 40-50%) of remaining severely disabled, a scenario called "futile recanalization". One of the causes for this lack of treatment effect is capillary obstruction, or "no reflow", potentially resulting from activated neutrophils and micrometer-sized blood clots. Previous work in rodent stroke models demonstrated that removal of these capillary stalls indeed improves reperfusion and recovery after stroke. However, there is a lack of knowledge regarding the role of neutrophils or microclots in patients with stroke, and their potential to indicate reperfusion failure.

Aim:

The goal of our study is to search for activated neutrophils and microclots in peripheral blood samples from patients with stroke. We anticipate that neutrophil and microclot characteristics such as size, shape, or surface structure may indicate stroke risk, and may be associated with clinical outcome, stroke ethology and reperfusion failure in patients with stroke. Our goal is to improve the prediction of stroke risk and treatment success.

Methodology:

We plan to prospectively include 500 patients with acute and chronic stroke, as well as a control group. We have teamed up with biophysicists from the Swiss Federal Laboratories for Materials Science (EMPA) using the novel microscopic tools 3D rotational digital tomography (DHTM) to achieve an unprecedented resolution of less than 10 μm for detection of altered neutrophil phenotypes and microclots in peripheral blood samples. Furthermore, in patients undergoing mechanical thrombectomy, retrieved clots will be analyzed with high-density micro-computertomography (micro-CT). Quantity, mechanical and structural properties of microclots and neutrophils will be correlated with risk of reperfusion failure, stroke recurrence and clinical recovery. Analyses of clots from patients with large vessel occlusion will be used to derive risk of reperfusion failure along with most likely source of the clot, and thus, most likely stroke etiology.

Potential Significance:

Current diagnostic tools are insufficient to predict response to treatment, clot source or stroke recurrence risk. Our project has the potential to discover new, clinically applicable biomarkers identifying patients at risk within a few hours, enabling individualized stroke treatment and prevention.

ELIGIBILITY:
Inclusion Criteria:

Patients without acute stroke CS or CSG

* No previous stroke or previous stroke ≥ 1 year ago
* Signed informed consent

Patients with acute stroke (AS-noTx, AS-IVT, AS-MT):

* Patients admitted with high suspicion of acute ischemic stroke
* Time of onset of stroke symptoms ≤ 12 hours
* Consent according to the regulations of research in an emergency situation
* Ischemic stroke later confirmed

Exclusion Criteria:

All groups:

* Pregnancy
* Age under 18 years

Acute Stroke no Therapy

• Acute treatment with IVT or with MT

Acute Stroke IVT-Group • Acute treatment with MT or without IVT

Acute Stroke MT-Group

• Acute treatment without MT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients without acute stroke (Control Group and chronic Stroke Group) will be recruited at the neurovascular ambulatory of the University Hospital Zurich
  Patient with acute stroke will be included at the stroke unit of the University Hospital Zurich.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Quantification and characterization of microclots | First Visit/Admission and patients with acute stroke after 24 hours, 3 months and 1 year
  3D rotational digital tomography and atomic force microscopy
  imaging outcome measurements:
  * size: length (µm), width (µm)
  * dry mass (g/dl)
  * praevalence (count in numbers)
  * composition (platelet aggregate vs. fibrin-rich microclots vs. microclot composite)
Quantification and characterization of neutrophils | First Visit/Admission and patients with acute stroke after 24 hours, 3 months and 1 year
  3D rotational digital tomography and atomic force microscopy
  image morphological outcome measurements:
  * size: diameter (µm), surface area (µm2), volume (fl), thickness (µm), sphericity
  * dry mass (g/dl)
  * praevalence (count in numbers)
  * activation state (activated vs. not activated vs. dead)
Evaluation of reperfusion failure in patients with large vessel occlusion and mechanical thrombectomy | <24 hours in patients with mechanical thrombectomy
  Defined by successfull macrovascular reperfusion (TICI >=2c) and insufficient microvascular reperfusion with the outcome measurment (yes/no)
  Successfull macrovasular reperfusion is defined according to the mTICI score 2c or 3.
  Microvascular reperfusion success will be evaluated with thresholds were used to discriminate between microvascular hypoperfusion and reperfusion, calculated from perfusion images obtained on computed tomography (CTP) or magnetic resonance perfusion imaging (MRP).

SECONDARY OUTCOMES:
Change in National Institute of Health Score Scale (NIHSS) | First Visit/Admission and patients with acute stroke after 24 hours, 3 months and 1 year
  will be assessed using National Institutes of Health Stroke Scale (NIHSS)
  NIHSS
  13 assessed functional domains Range 0-42, higher score indicates severe impairment
Degree of disability or dependence assessed by the modified ranking scale (mRS) | First Visit/Admission and patients with acute stroke after 24 hours, 3 months and 1 year
  will be assessed using modified Rankin Scale (mRS)
  mRS
  Range: (0-6) 0 = no symptoms, 6 = death, higher score indicates severe impairment
Assessment Quality of Life using European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) | 365 days
  EQ-5D-5L
  Evaluation of 5 different aspects of health with likert scale (1-5)
  MOBILITY SELF-CARE USUAL ACTIVITIES PAIN / DISCOMFORT ANXIETY / DEPRESSION Each domain is scored individually, higher values indicate higher impairment of quality of life
Incidence of new cardiovascular disease | 365 days
  Stroke, heart attack, brain bleeding
All-cause mortality | 365 days
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Wegener, Prof., Principal Investigator — University Hospital Zurich, department Neurology
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided upon reasonable request